CLINICAL TRIAL: NCT03448120
Title: Acupuncture and Dry Needling in Peripheral Acute Fatigue Reduction Induced in Biceps Brachialis: Cross-Sectional Study
Brief Title: Acupuncture and Dry Needling in Peripheral Acute Fatigue Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria das Graças Rodrigues de Araújo, Professor of the Physiotherapy Department, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Muscle Fatigue, Acupunture and; UFPE (Registry Identifier: CAAE N. 79139717.6.0000.5208)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Sedentary Lifestyle; Males
Keywords: Muscle fatigue; Thermography; Acupuncture; Dry needling
MeSH Terms: conditions — Sedentary Behavior | interventions — Acupuncture Therapy; Dry Needling

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): The volunteers who will remain in prolonged rest (10 minutes for homeostasis plus 30 minutes of no intervention).
- Acupuncture Group (Experimental): The volunteers will receive six needles in six acupoints in the non-dominant upper limb for 30 minutes.
  Interventions: Procedure: Acupuncture
- Dry needling Group (Experimental): The volunteers will receive application of six needles arranged in the non-dominant biceps brachialis for 30 minutes.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Acupuncture — Six needled will be inserted in six already defined acupoints along the non-dominant upper limb for a period of 30 minutes.
  Arms: Acupuncture Group
Procedure: Dry needling — Six needles will be inserted in six predefined points along the volunteers non-dominant biceps brachialis for 30 minutes.
  Arms: Dry needling Group

SUMMARY:
Introduction: Neuromuscular fatigue is defined when the muscle becomes incapable of generating muscle power or strength after exercise or long repetitive activities. As well as, the inability to maintain optimum performance and generate maximum voluntary contractions during a physical exercise. When performing physical activity, the body's metabolic response increases proportionally to exercise to satisfy the demands of the human physiological. Part of the energy accumulated during exercise is lost to the environment in the form of heat and another part is maintained internally through the physiological control for thermoregulation. In addition, the muscle generates an electric signal important to determine its status regarding power and fatigue.

Objective: To investigate the reduction of acute peripheral fatigue induced by isometric contractions from acupuncture and dry needling techniques, compared to absolute rest.

Methods: This is a cross-sectional study and experimental study, with descriptive, analytical and quantitative approach. It follows the Consolidated Standards of Reporting Trials (CONSORT) guidelines. The volunteers will be gathered according to the eligibility criteria, and randomly divided in 3 groups: the control group (G1), the volunteers who will remain in prolonged rest; the acupuncture group (G2), in which volunteers will receive six needles in six acupoints in the non-dominant upper limb and the dry needling group (G3), in which the volunteers will receive application of six needles arranged in the non-dominant biceps brachialis.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals, aged between 18 and 40 years and who are not practicing regular physical activity (sedentary lifestyle).

Exclusion Criteria:

* Are using food supplementation;
* Have joint or bone lesions on the limb to be studied;
* Have problems of metabolic order;
* Use of hormone therapy;
* Have had caffeine in the two hours before the study;
* Have ulceration or wounds in the electrode application region for electromyography;
* Show absence of myofascial trigger points in areas of dry needling technique;
* Body Mass Index below normal values or higher than overweight.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Perception of muscle fatigue | 60 minutes
  Fatigue perception measured by Visual Analog Scale for fatigue assessment, graduated from 0,00 to 10,0 centimeters, being 0,00 no fatigue and 10,0 maximum fatigue.
Muscle temperature | 60 minutes
  Infrared thermographic Imaging analysis of acute peripheral muscle fatigue.
Muscle fatigue | 60 minutes
  Electromyographic activity (in microvolts) of the biceps brachii muscle to assess muscle fatigue through the median frequency (MF).

OTHER OUTCOMES:
Contraction time | 60 minutes
  The time of intermittent isometric contractions was delimited by the number of valid contractions during each exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Kinesiotherapy and Manual Therapeutic Resources, Department of Physical Therapy, Federal University of Pernambuco (UFPE), Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Antonino GB, Paula de Lima Ferreira A, Nepomuceno Montenegro EJ, Galvao de Moura Filho A, Freire da Silva AF, de Araujo MDGR. Acupuncture and Dry Needling in the Reduction of Peripheral Acute Fatigue Induced in the Biceps Braquii: Protocol for a Single-blinded Randomized Controlled Clinical Trial. J Acupunct Meridian Stud. 2020 Oct;13(5):163-166. doi: 10.1016/j.jams.2020.08.001. Epub 2020 Sep 1. PMID 32889135